CLINICAL TRIAL: NCT07008755
Title: Clinical Trial of Different Doses of Pegylated Interferon α-2b Injection Nebulization Therapy for Common Hand, Foot, and Mouth Disease (HFMD).
Brief Title: Clinical Trial of Pegylated Interferon α-2b Via Nebulization for Treatment of Hand, Foot, and Mouth Disease .
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhengzhou Children's Hospital, China (Other)
Responsible Party: Principal Investigator, Fang Wang, Chief physician, Zhengzhou Children's Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC-C-007-A04
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: HFMD
Keywords: Peginterferon α-2b injection; HFMD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peginterferon α-2b 45 mcg dose group (Experimental)
  Interventions: Drug: Peginterferon α-2b injection
- Peginterferon α-2b 90 mcg dose group (Experimental)
  Interventions: Drug: Peginterferon α-2b injection

INTERVENTIONS:
Drug: Peginterferon α-2b injection — During the study period, patients will continue to receive symptomatic supportive therapy, along with nebulized Peginterferon α-2b injection at a dose of 45 μg per administration, to be delivered on Day 1 and Day 3.
  Arms: Peginterferon α-2b 45 mcg dose group
Drug: Peginterferon α-2b injection — CoDuring the study period, patients will continue to receive symptomatic supportive therapy, along with nebulized Peginterferon α-2b injection at a dose of 90 μg per administration, to be delivered on Day 1 and Day 3.
  Arms: Peginterferon α-2b 90 mcg dose group

SUMMARY:
This is a multicenter clinical trial investigating the safety and efficacy of inhaled Peginterferon α-2b at different doses, in combination with supportive care, for the treatment of patients with hand, foot, and mouth disease (HFMD) of ordinary type. The trial aims to enroll 90 patients with HFMD. Eligible subjects will be randomly assigned to receive either supportive care + Peginterferon α-2b mcg or supportive care + Peginterferon α-2b 90 mcg, administered on days 1 and 3. The study period includes a 3-day screening phase and a 5-7 day inpatient visit period. The results of this trial will be used to evaluate safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

-1. Age: 1 year of age ≤ Age ≤ 6 years of age. 2.Gender: Both male and female. 3.Clinical symptoms/signs: Manifesting as common type HFMD (Stage 1, rash stage), with fever or rash symptoms first occurring within 72 hours prior to the signing of the informed consent form.

4.Informed consent: Guardians understand and sign the informed consent form (if the guardian is the parent, both parents must sign).

Exclusion Criteria:

* (1) Severe or Critical HFMD Presentation at Enrollment

  1. Manifesting as severe HFMD (Stage 2, neurological involvement phase)
  2. Manifesting as critical HFMD (Stage 3 or 4, cardiopulmonary failure phase) with any of:

     Brainstem encephalitis, encephalomyelitis, or meningitis,Neurogenic pulmonary edema or respiratory failure requiring mechanical ventilation,Shock or circulatory collapse.
  3. Concurrent multi-organ failure requiring ICU monitoring

     (2) Allergy History and Treatment History

  <!-- -->

  1. Received interferon, ribavirin, acyclovir, ganciclovir, or vidarabine monophosphate within 30 days prior to screening or current use
  2. Received immunoglobulin or glucocorticoid therapy within 30 days prior to screening or current use
  3. Known hypersensitivity to interferon or its components, or other clinically significant allergies contraindicating participation
  4. Use of other investigational drugs within 3 months or 5 half-lives (whichever is longer) prior to screening, or current participation in medical device trials

     (3) Medical History

  <!-- -->

  1. Congenital heart disease, severe malnutrition, immune dysfunction, asthma, or other severe systemic diseases
  2. Active HBV, HCV, HIV, or Treponema pallidum infection
  3. History of malignant tumors (current or prior)
  4. History of epilepsy, neurological/psychiatric disorders, or relevant family history

     (4) Clinical Parameters: Resting respiratory rate >40 breaths/min,Heart rate >160 bpm

     (5) Other Considerations: Any condition deemed by investigators to render participation medically inadvisable

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Median time to resolution of fever | Day5-7.
Median time to resolution of skin rash | Day5-7.
Median time to resolution of oral ulcers | Day5-7.
Median time to resolution of feeding difficulties | Day5-7.

SECONDARY OUTCOMES:
Proportion of patients with complete recovery of fever | Day 3
Proportion of patients with complete recovery of fever | Day 5
Proportion of patients with complete recovery of rash | Day 3
Proportion of patients with complete recovery of rash | Day 5
Proportion of patients with complete recovery of oral ulcers | Day 3
Proportion of patients with complete recovery of oral ulcers | Day 5
Proportion of patients with complete recovery of feeding difficulties | Day 3
Proportion of patients with complete recovery of feeding difficulties | Day 5
Proportion of patients showing improvement in fever | Day 3
Proportion of patients showing improvement in fever | Day 5
Proportion of patients showing improvement in rash | Day 3
Proportion of patients showing improvement in rash | Day 5
Proportion of patients showing improvement in oral ulcers | Day 3
Proportion of patients showing improvement in oral ulcers | Day 5
Proportion of patients showing improvement in feeding difficulties | Day 3
Proportion of patients showing improvement in feeding difficulties | Day 5
Proportion of patients developing pulmonary edema | Day1-7
Proportion of patients developing myocarditis | Day1-7
Proportion of patients developing respiratory failure | Day1-7
Proportion of patients developing circulatory failure | Day1-7
Proportion of patients developing meningoencephalitis | Day1-7
Proportion of patients achieving viral nucleic acid negativity | Day 3
Proportion of patients achieving viral nucleic acid negativity | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Fang Wang, Principal Investigator — Henan Children's Hospital Zhengzhou Children's Hospital
Locations (5):
- China (5):
  - Xindu District People's Hospital of Chengdu, Chengdu
  - The Seventh People's Hospital of Liangshan Yi Autonomous Prefecture, Liangshan
  - Henan Children's Hospital (Zhengzhou Children's Hospital), Zhengzhou
  - Zhengzhou People's Hospital, Zhengzhou
  - Ziyang Central Hospital, Ziyang